CLINICAL TRIAL: NCT06400394
Title: Impact of Surgical Site Infection in Peritonitis After Peritoneal Lavage With Super-oxidixed Solution: A Randomised Double-Blind, Placebo-controlled Trial
Brief Title: Impact of Surgical Site Infection in Peritonitis After Peritoneal Lavage With Super-oxidixed Solution
Acronym: Plasso 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Hospital Queen Elizabeth, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dinesh Alagoo, Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSCH ID-24-01241-VGD
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Surgical Site Infection
Keywords: "Peritonitis" "Peritoneal lavage" "surgical site infection" "super-oxidised solution"
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: a randomised double blind placebo controlled parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: computerized block randomization using the website www.randomization.com with a block size of 8 and allocation ratio of 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Peritoneal lavage with normal saline 0.9% 1L and wound lavage with normal saline 0.9% 500ml
  Interventions: Device: Normal Saline
- Study group (Experimental): Peritoneal lavage with super-oxidised solution of at least 1L and wound lavage with super-oxidised solution of 500ml
  Interventions: Device: Hydrocyn Aqua®

INTERVENTIONS:
Device: Hydrocyn Aqua® — The study solution comes in a liquid form containing hypochlorous acid (HOCl) in a concentration of 0.003%. It is used as a topical agent for wound and peritoneal lavage before wound closure
  Arms: Study group
Device: Normal Saline — aqueous solution of electrolytes and other hydrophilic molecules
  Arms: Control group

SUMMARY:
This is randomised double blinded placebo-controlled parallel-group study. Patients in Hospital Queen Elizabeth, Sabah and Hospital Universiti Sains Malaysia, Kelantan who undergo laparotomy for peritonitis will be equally randomised into two groups : intervention group receiving super-oxidised solution and the control group receiving normal saline during peritoneal and wound lavage.

This is a superiority study assessing the effectiveness of the intervention. The patient and doctors directly involved in the partient care will be blinded in this study

DETAILED DESCRIPTION:
OBJECTIVES

PrimaryOutcome:

To evaluate the effectiveness of peritoneal lavage with superoxidised solution in reducing incidence of surgical site infection after open surgery for peritonitis.

SecondaryOutcome:

i.To evaluate the effectiveness of peritoneal lavage with super-oxidised solution in reducing inflammatory markers C-reactive protein(CRP) at 24 and 48 hours after open surgery for peritonitis ii.To evaluate the effectiveness of peritoneal lavage with super oxidised solution in reducing duration of post-operative ileus after open surgery for peritonitis.

METHODOLOGY

Study Design This is a randomised double blind placebo controlled parallel group study. This is a superiority study assessing the effectiveness of the intervention. The patients and doctors directly involved in the patient care will be blinded in this study.

Masking Study participants were randomly assigned following computerized block randomization using the website www.randomization.com with a block size of 8 and allocation ratio of 1:1. Allocation sequence and concealment will be performed by the research staff from the Clinical Research Centre who had no clinical involvement in the trial. The allocation sequence will be concealed from the researcher enrolling and assessing the participants in sequentially numbered, opaque, sealed envelopes.

The study participants, healthcare providers who attend to the participants during the trial (surgeon and nurses), outcome evaluators (surgical doctors and nurses) and data collectors will be blinded to the allocation.

2 arms with 56 participants per arm Study group: Peritoneal lavage with super-oxidised solution of at least 1L and wound lavage with super-oxidised solution of 500ml [Super-oxidised solution used in this study is Hydrocyn Aqua® (Vigilenz MD., Penang, Malaysia)] Control group: Peritoneal lavage with normal saline 0.9% 1L and wound lavage with normal saline 0.9% 500ml

Enrollment The estimated total number of participants to be enrolled is about 116 with 20% dropout rate

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 13yrs and above
2. Diagnosed with perforated viscus intraoperatively
3. Undergo Midline Laparotomy
4. ASA 3 and below

Exclusion Criteria:

1. Surgical technique: Laparoscopic washouts
2. Patients on steroid treatment and immunosuppressant therapy.
3. More than ASA 3
4. Inability to give/understand informed consent
5. Revision-surgery (previous abdominal surgery within the last 30 days)
6. Planned re-laparotomy within 30 days
7. Terminal kidney failure requiring dialysis
8. Concurrent abdominal wall infections

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
SSI Incidence | 30 days
  To evaluate the effectiveness of peritoneal lavage with superoxidised solution in reducing incidence of surgical site infection after open surgery for perforated viscus.

SECONDARY OUTCOMES:
CRP Level | 24-48 hrs
  To evaluate the effectiveness of peritoneal lavage with super-oxidised solution in reducing inflammatory markers C-reactive protein(CRP) at 24 and 48 hours after open surgery for perforated viscus
Flatus time | 1-2 days
  To evaluate the effectiveness of peritoneal lavage with super oxidised solution in reducing duration of post-operative ileus after open surgery for perforated viscus.